CLINICAL TRIAL: NCT02291341
Title: Single Dose Crossover Comparative Bioavailability Study of Duloxetine Delayed-Release Capsules 60 mg in Healthy Adult Human Subjects Under Fed Conditions
Brief Title: Bioavailability Study of Duloxetine Delayed-Relase Capsules 60 mg Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BA0859089-01
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2008-07

CONDITIONS: Healthy
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Duloxetine Delayed-Release Capsules, 60 mg (Experimental): Duloxetine Delayed-Release Capsules, 60 mg of Dr. Reddys Laboratories Limited
  Interventions: Drug: Duloxetine
- Cymbalta (Active Comparator): Cymbalta® 60 mg capsule of Eli Lilly and Company
  Interventions: Drug: Cymbalta®

INTERVENTIONS:
Drug: Duloxetine — Duloxetine Delayed-Release Capsules 60 mg
  Other Names: Cymbalta
  Arms: Duloxetine Delayed-Release Capsules, 60 mg
Drug: Cymbalta® — 60 mg capsule of Eli Lilly and Company
  Arms: Cymbalta

SUMMARY:
This study were to compare the relative bioavailability of Duloxetine HCl delayed release capsule 60 mg with that of 'CYMBALTA®' delayed release capsule 60 mg (Duloxetine HCl delayed release capsule 60 mg) in healthy, adult, human subjects under fed conditions and to monitor safety of subjects

DETAILED DESCRIPTION:
Open label, randomized, two period, two treatment, two sequence, crossover, balanced, single dose comparative oral bioavailability study in healthy, adult, human subjects under fed conditions

ELIGIBILITY:
Inclusion Criteria:

1. The subjects should be healthy human between 18 and 45 years.
2. The subjects should be screened within 21 days prior to the administration of first dose of the study drug.
3. The subjects should have a BMI between 18.5 and 24.9 weight in kg/ height2 in meter.
4. The subjects should be able to communicate effectively with study personnel.
5. The subjects should be able to give written informed consent to participate in the study.

   If subject is a female volunteer and
6. Is of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence.
7. Is postmenopausal for at least 1 year.
8. Is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject).

Exclusion Criteria:

1. The subjects who have a history of allergic responses to Duloxetine or other related drugs.
2. The subjects who have significant diseases or clinically significant abnormal findings during screening, medical history, physical examination, laboratory evaluations, ECG and X-ray recordings.
3. The subjects who have any disease or condition which might compromise the haemopoeitic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system, diabetes, psychosis or any other body system.
4. The subjects who have a history or presence of bronchial asthma.
5. The subject who have used enzyme-modifying drugs within 30 days prior to receiving the first dose of study medication.
6. The subjects who have history of drug dependence, recent history of alcoholism or of moderate alcohol use.
7. The subjects who are smokers, who smoke more than or equal to 10 cigarettes per day or more than or equal to 20 biddies per day or those who cannot refrain from smoking during study period.
8. The subjects with a history of difficulty with donating blood or difficulty in accessibility of veins.
9. The subjects who have donated (1 unit: 350 ml / 450 ml) blood within 90 days prior to receiving the first dose of study medication.
10. The subjects who have a positive hepatitis screen (includes subtypes A, B, C & E).
11. The subjects who have a positive test result for HIV antibody and / or syphilis (RPR/VDRL).
12. The subject who receives an investigational product, or has participated in a drug research study within a period of 90 days prior to the first dose of the study medication administration.
13. Female volunteers demonstrating a positive pregnancy screen.
14. Female volunteers who are currently breast-feeding.
15. Female volunteers not willing to use contraception during the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2008-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) | 1.0, 2.0,3.0, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 9.0, 10.0, 11.0, 12.0, 24.0, 36.0, 48.0,60.0 and 72.0 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Ronak Modi, MBBS, Principal Investigator — BA Research India Ltd
Locations (1):
- BA Research India Ltd, Ahmedabad, Gujarat, India